CLINICAL TRIAL: NCT00376142
Title: Translating Clinicians' Beliefs Into Implementation Interventions (TRACII): a Modelling Experiment to Change Clinicians' Intentions to Implement Evidence-Based Practice.
Brief Title: Translating Clinicians' Beliefs Into Implementation Interventions (TRACII)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Newcastle University (Other)
Collaborators: Newcastle Primary Care Trust (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: TIME2005; QLRT-2001-00657
Record Dates: First submitted 2006-09-13; First posted 2006-09-14 (Estimated); Last update posted 2006-09-14 (Estimated); Status verified 2006-09

CONDITIONS: Upper Respiratory Tract Infection; URTI
Keywords: Intention; Behaviour; Evidence-based practice; Intervention
MeSH Terms: conditions — Respiratory Tract Infections; Behavior

INTERVENTIONS:
Behavioral: Psychological theory-based behaviour change interventions

SUMMARY:
Using a theory-based approach, the purpose of this study is to identify modifiable factors underlying professional behaviour in order to identify those processes to target with an implementation intervention and to gain an understanding of how interventions might work and thus be optimised.

Our principal objective is to develop interventions to change beliefs that have already been identified as antecedents to antibiotic prescribing for sore throats and then to experimentally evaluate these interventions to identify those which have the largest impact on behavioural intention

DETAILED DESCRIPTION:
It is a consistent finding that changing clinical practice is unpredictable and can be a slow and haphazard process. Over the last decade a considerable body of literature has been reviewed suggesting that a range of interventions (e.g. reminder systems, interactive education) can be effective in changing health care professionals' behaviour. However, studies have substantial heterogeneity of interventions used, targeted behaviours, and study settings that make generalising their findings to routine healthcare settings problematic - there is no underlying generalisable taxonomy for either research or service settings by which to characterise individuals, settings and interventions. The assumption that clinical practice is a form of human behaviour and can be described in terms of general theories relating to human behaviour offers the basis for a taxonomy for Implementation Research. For example, the effectiveness of interventions may be influenced by factors such as health professionals' beliefs or perceived control over their practice - generalisable concepts that can be used across different contexts. Two steps are necessary to design a theory-based intervention for a behaviour change trial: Step 1) The identification of modifiable factors underlying professional behaviour in order to identify those processes to target with an intervention (process modelling) Step 2) To gain an understanding of how interventions might work and thus be optimised (intervention modelling).

Our previous work has focussed on Step 1. The next step is to develop interventions to change beliefs based on identified theoretical predictors, and this is the focus of the present study. We will develop interventions to change the salient beliefs distinguishing high and low intenders, using previously identified GPs salient beliefs that predict their intention to prescribe antibiotics for patients with uncomplicated sore throat.

Design Theoretical framework: Theory of Planned Behaviour Methods: Postal questionnaire survey Clinical behaviour: Prescribing antibiotics for uncomplicated sore throat Participants: General Practitioners We will develop a sampling frame from lists of general practitioners supplied by Primary Care Groups in the North East of England. We will then sample to recruit sufficient general practitioners for the sample size of the experiments.

Previous work by the applicants has identified the salient beliefs of GPs that distinguish between those who intend to prescribe antibiotics and those who do not. Based on this information (and on-going work to produce a taxonomy of clinical behaviours and potential psychological behavioural technologies)we will select and develop two interventions designed to address changing the discriminative beliefs in the prescribing of antibiotics for sore throat.

The interventions will be evaluated in a three arm randomised controlled trial embedded in a questionnaire survey, using postal methods. The questionnaire package will be administered on two occasions.

For each administration of the questionnaire package, two reminders will be mailed to non-responding clinicians. In the light of our experience of the response rate in our previous study we plan to offer a £10 incentive to each subject to increase response rates. Subjects will receive a letter of invitation, and a study package that will include: a set instructions, an individually packaged set of materials for measuring behavioural simulation (patient scenarios), behavioural intention and process measures(Questionnaire) which they will be asked to read in this order. On the second administration the package will also contain the intervention, which GPs will be asked to open prior to completing the outcome and process measures.

ELIGIBILITY:
Inclusion Criteria:

* General Practitioner registered with a practice in the target Primary Care Trusts

Exclusion Criteria:

* None

Min Age: 0 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1200
Dates: Start 2005-04; Study Completion 2005-11

PRIMARY OUTCOMES:
Behavioural intention to prescribe antibiotics
Behavioural simulation (prescribing behaviour)

SECONDARY OUTCOMES:
Process measurement pre-intervention
Process measurement post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Martin P Eccles, MD, FMedSci, Principal Investigator — University of Newcastle Upon-Tyne
Locations (1):
- Institute of Health and Society, Newcastle University, Newcastle upon Tyne, United Kingdom

REFERENCES:
- [Derived] Hrisos S, Eccles M, Johnston M, Francis J, Kaner EF, Steen N, Grimshaw J. Developing the content of two behavioural interventions: using theory-based interventions to promote GP management of upper respiratory tract infection without prescribing antibiotics #1. BMC Health Serv Res. 2008 Jan 14;8:11. doi: 10.1186/1472-6963-8-11. PMID 18194527
- [Derived] Hrisos S, Eccles M, Johnston M, Francis J, Kaner EF, Steen N, Grimshaw J. An intervention modelling experiment to change GPs' intentions to implement evidence-based practice: using theory-based interventions to promote GP management of upper respiratory tract infection without prescribing antibiotics #2. BMC Health Serv Res. 2008 Jan 14;8:10. doi: 10.1186/1472-6963-8-10. PMID 18194526